CLINICAL TRIAL: NCT04543370
Title: A Phase 1, Open-Label Study to Evaluate CYP3A4 Drug-Drug Interactions of Edasalonexent in Healthy Adult Subjects
Brief Title: Study of Edasalonexent With Midazolam and Deflazacort in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CAT-1004-106
Record Dates: First submitted 2020-08-21; First posted 2020-09-10 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — edasalonexent; Midazolam; deflazacort

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): 2 mg midazolam on Day 1 and 36 mg deflazacort on Day 2.
  Interventions: Drug: Midazolam 2 MG/ML; Drug: Deflazacort 36Mg Tab
- Treatment B (Experimental): 2000 mg edasalonexent TID on Day 1 to Day 11 with 2 mg midazolam on Day 10 and with 36 mg deflazacort on Day 11.
  Interventions: Drug: Edasalonexent 2000 mg TID; Drug: Midazolam 2 MG/ML; Drug: Deflazacort 36Mg Tab

INTERVENTIONS:
Drug: Edasalonexent 2000 mg TID — CAT-1004 capsules
  Arms: Treatment B
Drug: Midazolam 2 MG/ML — 2 mg/ml syrup
Drug: Deflazacort 36Mg Tab — 36 mg tablets

SUMMARY:
Drug-drug interaction (DDI) and Cardiodynamic Evaluation Study To assess the effect of multiple oral doses of edasalonexent on the single-dose pharmacokinetics (PK) of midazolam (a cytochrome P450 [CYP]3A4 sensitive substrate) and of deflazacort (a CYP3A4 moderate sensitive substrate) in healthy adult subjects.

DETAILED DESCRIPTION:
This is an open-label, fixed-sequence DDI and cardiodynamic study in healthy adult subjects.

Twenty-six (26), healthy, adult male and female (non-childbearing potential) subjects will be enrolled.

Screening of subjects will occur within 28 days prior to the first dosing.

To assess the effect of multiple oral doses of edasalonexent on the single-dose pharmacokinetics (PK) of midazolam (a cytochrome P450 [CYP]3A4 sensitive substrate) and of deflazacort (a CYP3A4 moderate sensitive substrate) in healthy adult subjects.

Visit assessments include Clinical laboratory tests, Safety ECGs and Cardiodynamic ECGs. Subjects will be housed on Day -3 of Period 1, until after the 24-hour blood draw and/or study procedures are completed on Day 12 of Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female (of non-childbearing potential), 18-55 years of age, inclusive at Screening
* Non-smoker
* Body mass index (BMI) ≥18.0 and ≤32.0 kg/m2 at Screening
* Medically healthy with no clinically significant medical history
* Ability to swallow multiple capsules/tablets.
* Ability to understand the study procedures, willing and able to comply with the protocol

Exclusion Criteria:

* History or presence of clinically significant medical condition or disease
* History or presence of hypersensitivity to edasalonexent or excipients based upon known allergies to compounds of a similar class such as salicylates, fish oil, eicosapentaenoic acid, or DHA
* History or presence of hypersensitivity to midazolam, deflazacort, or related compounds (e.g., steroids or their formulation including lactose).
* Participation in another clinical study within 30 days prior to the first dosing

Ages: 18 Years to 55 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2020-09-06 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
AUC of edasalonexent with midazolam and deflazacort | 12 Days

SECONDARY OUTCOMES:
QTc interval with edasalonexent | 12 Days
Number of participants with reported treatment-related adverse events | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Donovan, MD, PhD, Study Chair — Chief Medical Officer, Catabasis
Locations (1):
- Celerion Clinical Research Unit, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No